CLINICAL TRIAL: NCT00791102
Title: A Randomized, Double-Blind, Placebo-Controlled, Cross-Over Trial of Topical ASP-1001 (Contrast Media Formulation) in the Prevention of the Signs and Symptoms of the Acute Response to Nasal Allergen Challenge (NAC)
Brief Title: Topical ASP-1001 (Contrast Media Formulation) and the Acute Response to Nasal Allergen Challenge (NAC)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Asphelia Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Robert Naclerio, Professor, University of Chicago
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 16504B (ASP2002-AR-01)
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Topical ASP-1001
  Interventions: Drug: ASP-1001 nasal spray
- 2 (Placebo Comparator): Placebo for Topical ASP-1001
  Interventions: Drug: Placebo for ASP-1001

INTERVENTIONS:
Drug: ASP-1001 nasal spray — 2 sprays (total 200 microliters) in each nostril 20 minutes before allergen challenge.
  Arms: 1
Drug: Placebo for ASP-1001 — 2 sprays (total 200 microliters) in each nostril 20 minutes before allergen challenge.
  Arms: 2

SUMMARY:
The purpose of this study is to see whether ASP-1001 when given as a nasal spray is safe and can reduce the signs and symptoms of allergic rhinitis (hayfever) following nasal challenge with antigen.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 55 years of age.
2. History of grass and/or ragweed allergic rhinitis.
3. Positive skin test to grass and/or ragweed antigen.
4. Positive response to screening nasal challenge.

Exclusion Criteria:

1. Physical signs or symptoms suggestive of renal, hepatic or cardiovascular disease.
2. Pregnant or lactating women.
3. Upper respiratory infection or sinusitis within 14 days of study start.
4. Use of nasal steroids, antihistamines in the last 2 weeks.
5. FEV1<80% of predicted at screening for subjects with history of mild asthma
6. current smokers or recent ex-smokers
7. Any social or medical condition that, in the opinion of the investigator, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Days to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical ASP-1001: Topical ASP-1001
  ASP-1001 nasal spray : 2 sprays (total 200 microliters) in each nostril 20 minutes before allergen challenge.
- Placebo for Topical ASP-1001: Placebo for Topical ASP-1001
  Placebo for ASP-1001 : 2 sprays (total 200 microliters) in each nostril 20 minutes before allergen challenge.
Period: Period 1
Arm/Group | Topical ASP-1001 | Placebo for Topical ASP-1001
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout Period of 2 Weeks
Arm/Group | Topical ASP-1001 | Placebo for Topical ASP-1001
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Topical ASP-1001 | Placebo for Topical ASP-1001
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 33 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Sneezing Symptom
Description: Sneezes. The change is calculated by adding the number of sneezes following both antigen challenges minus twice the number of sneezes after the diluent challenge.
Time Frame: 10 minutes after diluent challenge and 10 minutes after each antigen challenge
Measure: Median (Inter-Quartile Range); unit: sneezes
Arm/Group | Topical ASP-1001 | Placebo for Topical ASP-1001
Number analyzed (Participants) | 20 | 20
sneezes | 1 [0 to 2] | 1 [0 to 8]

2. Secondary Outcome: Nasal Peak Inspiratory Flow Measurements
Description: The value of nasal peak inspiratory flow. The change is calculated by adding the values of nasal peak inspiratory flow following both antigen challenges minus twice the value of nasal peak inspiratory flow after the diluent challenge.
Time Frame: 15 minutes after diluent challenge and 15 minutes after each antigen challenge
Measure: Median (Inter-Quartile Range); unit: L/min
Arm/Group | Topical ASP-1001 | Placebo for Topical ASP-1001
Number analyzed (Participants) | 20 | 20
L/min | -8.5 [-51.25 to 3.75] | -30 [-40 to -20]

3. Primary Outcome: Change in Runny Nose Symptom
Description: The nasal symptoms on a scale of 0-3 (0=no symptoms, 1=mild, 2= moderate, 3= severe). The change is calculated by adding the score of runny nose following both antigen challenges minus twice the score of runny nose after the diluent challenge.
Time Frame: 10 minutes after diluent challenge and 10 minutes after each antigen challenge
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Topical ASP-1001 | Placebo for Topical ASP-1001
Number analyzed (Participants) | 20 | 20
units on a scale | 1 [0 to 3] | 2.5 [0 to 4]

4. Primary Outcome: Change in Stuffy Nose Symptom
Description: The nasal symptoms on a scale of 0-3 (0=no symptoms, 1=mild, 2= moderate, 3= severe). The change is calculated by adding the score of stuffy nose following both antigen challenges minus twice the score of stuffy nose after the diluent challenge.
Time Frame: 10 minutes after diluent challenge and 10 minutes after each antigen challenge
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Topical ASP-1001 | Placebo for Topical ASP-1001
Number analyzed (Participants) | 20 | 20
units on a scale | 1 [0 to 2.75] | 2 [0.25 to 3]

5. Primary Outcome: Change in Itching Symptom
Description: The nasal symptoms on a scale of 0-3 (0=no symptoms, 1=mild, 2= moderate, 3= severe). The change is calculated by adding the score of itchy nose following both antigen challenges minus twice the score of itchy nose after the diluent challenge.
Time Frame: 10 minutes after diluent challenge and 10 minutes after each antigen challenge
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Topical ASP-1001 | Placebo for Topical ASP-1001
Number analyzed (Participants) | 20 | 20
units on a scale | 0 [0 to 2.75] | 1 [0 to 2]

6. Secondary Outcome: Change in Nasal Peak Inspiratory Flow Measurements From Before to After Treatment
Time Frame: 15 minutes prior to treatment and 15 minutes post antigen challenges
Measure: Median (Inter-Quartile Range); unit: L/min
Arm/Group | Topical ASP-1001 | Placebo for Topical ASP-1001
Number analyzed (Participants) | 20 | 20
L/min | -7.5 [-20 to 0] | -10 [-20 to 9.5]

ADVERSE EVENTS:
Arm/Group | Topical ASP-1001 | Placebo for Topical ASP-1001
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No